CLINICAL TRIAL: NCT03223506
Title: Validation of a Physiological Based Pharmacokinetic Model by the Study of Paracetamol Distribution in the Brain Compartments in Brain Injured Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PB-PK BRAIN
Record Dates: First submitted 2017-05-22; First posted 2017-07-21 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2017-10

CONDITIONS: Brain Injured Patients
MeSH Terms: interventions — Acetaminophen

ARMS (1):
- Paracetamol arm (Experimental): Administration of 10 mg/ml of paracetamol
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Drug: Paracetamol

SUMMARY:
Brain is composed of several anatomical compartments separated by physiological barriers allowing the maintenance of homeostasis. Furthermore, brain-barriers restrain the diffusion of some drugs in cerebro spinal fluid (CSF) and in extracellular fluid (ECF) of brain tissue, making the development and optimization of dosing regimen of new drugs difficult. Most dosing regimen are determined from the plasma concentration because target site concentrations are difficult to obtain in the brain, hence making the prediction of the therapeutic effect, the adverse effect and the toxicity of a brain- diffused drug difficult. Although quantitative and qualitative differences exist in the processes governing pharmacokinetic (PK) in CSF and brain tissue, CSF is considered as the best surrogate of drugs penetration in the human brain.

A study previously published has evaluated in rats the cerebral distribution of paracetamol, used as a marker of passive diffusion in the ECF by microdialysis in the striatum and in the CSF by microdialysis in the ventricular lateralis and the cistern magna. Authors chose paracetamol, as it has the property to diffuse passively and rapidly in the central nervous system allowing the exclusive description of the relationship between the different compartments of the brain. This study has first revealed an unexpected important difference between the distribution profiles obtained in ECF and CSF. Based on these results, authors developed a physiologically based PK model (PBPK) to describe their results and thereby offering the possibility to perform interspecies simulations to predict central nervous system (CNS) distribution of paracetamol in human. In this study, authors used this model to perform pharmaceutical extrapolations between species converting data from animal to human by replacing obtained data from clinical past studies describing paracetamol distribution in the CSF and in plasma.

Microdialysis allows determination of free extracellular concentrations of drug in different tissues and also in brain. Our research team, INSERM U1070, has several past experiences with studies involving micro-dialysis to study the distribution of antibiotic in tissue in both animal and human including cerebral tissue in rat and human. Recommendation from the scholar society suggests that brain injured patients should benefit from a multimodal monitoring to optimize their care and brain perfusion. This invasive multimodal monitoring consists of measuring the intracranial pressure, the oxygen tissue-pressure, the estimation of the cerebral blood flow-rate by cranial Doppler as well as the monitoring of cerebral ischemic parameters by microdialysis. We also prevent systemic cerebral aggression among which, hyperthermia, explaining the prescription of paracetamol among a large number of brain injured patients. Furthermore setting up of an external ventricular draining (EVD) to treat an intra cranial hypertension is usually necessary to allow the continuous flow of the excess of CSF in the brain ventricle.

Few studies carried on human has aimed at comparing the distribution of drugs in both the CSF and the brain extracellular fluid though it is established that the brain barriers differ in their permeability as well as the drug's concentrations are different between brain compartments. Thus by mean of monitoring through microdialysis and/or through therapeutic EVD, required by brain-injured patients, we aim in our study to explore the pharmacokinetic of paracetamol in the brain ECF, the CSF and the plasma and to validate in man the PBPK developed in rat.

ELIGIBILITY:
Inclusion Criteria:

* Brain injured patient
* Age ≥ 18 ans
* Patient with a brain microdialysis monitoring and/or an external ventricular drainage
* Patient receiving paracetamol for clinical purpose

Exclusion Criteria:

* Paracetamol allergy
* Liver failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-03-23 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Area under the curve of paracetamol in the CSF, ECF and plasma. | 24 months

SECONDARY OUTCOMES:
Area under the curve ratio of plasmatic of paracetamol between 2 administrations | 30 months
Area under the curve ratio of free cerebral concentration (CSF and ECF) of paracetamol between 2 administrations | 30 months
Maximum concentration of paracetamol in cerebro spinal fluid | 30 months
Maximum concentration of paracetamol in extra cellular fluid | 30 months
Minimum concentration of paracetamol in cerebro spinal fluid | 30 months
Minimum concentration of paracetamol in extra cellular fluid | 30 months
Elimination half life of paracetamol in cerebro spinal fluid | 30 months
Elimination half life of paracetamol in extra cellular fluid | 30 months
Minimum plasma concentration | 30 months
Volume of distribution | 30 months
Clearance of paracetamol | 30 months
Maximum plasma concentration | 30 months
Elimination half life of paracetamol | 30 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Poitiers, Poitiers, France